CLINICAL TRIAL: NCT00299338
Title: A Pharmacokinetic and Safety Study of Procaine HCl in HIV-1 Infected Patients
Brief Title: A Dose Response and Safety Study of Procaine HCl in HIV-Infected Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Samaritan Pharmaceuticals, Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP01A-SII-101
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Last update posted 2006-04-03 (Estimated); Status verified 2006-03

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; CD4; HAART; antiretroviral; treatment failure; resistance; CCR4; CXCR5; gp120; gp41; cholesterol; lipid rafts; intracellular fluid; receptors; chemokine; antigens; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Drug: SP01A

SUMMARY:
This a Phase I/II non-randomized, open-label clinical study of 8 weeks duration using SP01A in HIV positive patients on a stable antiretroviral regimen. Dose response and safety associated with oral administration of four doses (200 mg, 400 mg, 600 mg, and 800 mg daily) of SP01A will be studied in a total of 24 study subjects. In addition, six HIV-negative subjects will be recruited as a control for cortisol secretion only and will not receive study medication.

DETAILED DESCRIPTION:
STUDY PLAN: DESCRIPTION This investigation will be a non-randomized, open-label study of four doses of SP01A in 24 individuals infected with HIV who are being treated with triple combination antiretroviral therapy. Additionally, a group of six HIV-negative subjects (group E) is being recruited as a control for cortisol secretion. This group will not receive study medication nor will they be evaluated for dose response or safety parameters.

DISCUSSION OF STUDY DESIGN, INCLUDING CONTROL GROUP Patients will receive the following doses of SP01A and will be divided into a low dose and high dose group for further analyses. There will be two segments within the low dose group. Group A will receive 200 mg of SP01A once per day. Group B will be administered 200 mg of SP01A twice daily. Similarly, there will be two segments in the high dose group. Group C will be treated with 200 mg of SP01A three times per day, while Group D will be administered 400 mg of SP01A twice daily.

A fifth group will also be introduced. This group, Group E, will serve as a control group and not receive any treatment.

The study will be conducted at a single investigative center (AIDS ReSearch Alliance, West Hollywood, CA). Six subjects with a diagnosis of HIV who are also receiving triple combination antiretroviral therapy and have been so doing for a minimum of 2 months are planned per group. Patients will be admitted to an in-patient facility for 72 hours. After an initial night to acclimate the patients to the facility, a 24-hour measurement of cortisol secretion in blood and urine will be conducted. After this is complete, patients will receive an initial single dose of SP01A orally. (200 mg SP-01A for group A, 400 mg for group B, 600 mg for group C, and 800 mg for group D). Blood and urine samples will also be collected for 24 hours to further evaluate the safety of the study medication. Patients will then be discharged from the facility.

After a 4-day washout, patients will return to the facility to start an 8-week dose-response study, sequentially using the four doses that will now be divided (200 mg daily for group A, 200 mg twice a day for group B, 200 mg three times per day for group C, and 400 mg twice daily for group D).

Subjects will return to the study center the day they are screened and as close to the same day of the week as practical during Weeks 1 (baseline), 2, 3, 4, 5, 6, 7, 8 (end of treatment) and 10 (post-treatment for examinations and specimen collection, as well as evaluation of reactions to study treatment). At the end of the 8-week drug administration period, patients will again be admitted to an in-patient facility for 72 hours. As before, patients will have an initial night to acclimate to the facility, followed by a 24-hour measurement of cortisol secretion in blood and urine. In the morning, following and ending the 24 hour basal cortisol secretion, patients in the four successive groups (A, B, C, and D), will receive their last dose of medication. They will also give their last blood and urine samples over the next 24 hours for additional safety sample collection. The total duration of study subject participation will be 11 weeks.

The six HIV negative subjects will be enrolled in group E. After an initial night to acclimate to the facility, blood and urine samples will be collected to determine baseline 24 hour blood and urine cortisol secretion. Patients will then be discharged. No study medication will be given to patients in group E.

ELIGIBILITY:
Inclusion Criteria:

1. Eighteen years of age or older (male or female).
2. If female, agreed to use suitable contraception to prevent pregnancy.
3. HIV positive as confirmed by viral load using nucleic acid sequence based amplification (NASBA), or enzyme-linked immunosorbent assay (ELISA) and Western Blot, for cohort A, B, C, and D. HIV negative by ELISA and Western blot for cohort E.
4. Karnofsky Performance Status score of at least 60.
5. No active opportunistic infection. Prophylaxis for MAl, CMV, Pneumocystis Pneumonia except Bactrim), or herpes was permitted.
6. Current CD4 count >200.
7. Stable triple therapy antiretroviral regimen (cohorts A, B, C, and D) for the preceding 8 weeks and willing to make no changes in regimen during the study.
8. Not taking any unapproved or experimental treatment for HIV, including antiretrovirals and immune modulators (such as interferons or interleukins).
9. Capable and willing to provide informed consent.
10. Agreed not to take Epoetin during the trial.
11. Baseline laboratory values:

Neutrophils > 1000 cells/mm3; Platelets > 75,000 cells/mL; SGOT <3 times upper limit of normal; SGPT <3 times upper limit of normal; Creatinine <2.0 mg/dL.

Exclusion Criteria:

1. Known or suspected allergy to procaine hydrochloride.
2. Patients taking DHEA supplementation or oral ketoconazole (which have anticortisol properties).
3. Patients using sulfonamides (including Septra/Bactrim).
4. Required use of sulfonamides, eg, Septra/Bactrim. (Procaine hydrochloride may inactivate sulfonamides).
5. Patients with glaucoma using anti-cholinesterase inhibitors (Humorsol [demecarium bromide] echothiophate iodide, Floropryl [isoflurophate], Isopto-Eserine [physostigmine salicylate]). Anti-cholinesterase Inhibitors should not be used while on procaine hydrochloride, since procaine itself has some anti-cholinesterase activity.
6. Patients with less than 6 months life expectancy.
7. Patients with adrenal insufficiency (determined by screening ACTH stimulation test).
8. Patients with lymphoma.
9. Patients with active hepatitis (viral or drug induced).
10. Patients with cancer, except peripheral Kaposi's sarcoma.
11. Patients on dialysis.
12. Patients who are pregnant.
13. Female patients of childbearing age who can not use two forms of birth control or abstain from sexual intercourse during the trial.
14. Any medical, psychological, psychiatric, or substance use problem that, in the opinion of the Principal Investigator, interferes with the patient's ability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 1997-09; Study Completion 2001-09

PRIMARY OUTCOMES:
Mean viral load reduction (log10) over 8 weeks
Maximal viral load suppression (LDL <50 & 400) over 8 weeks
Cortisol reduction over 8 weeks

SECONDARY OUTCOMES:
Improvement in quality of life indices (Whalen Scale) over 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Brown, MD, Principal Investigator — AIDS Research Alliance of West Hollywood
Locations (1):
- AIDS Research Alliance of West Hollywood, West Hollywood, California, United States